CLINICAL TRIAL: NCT04753320
Title: Remote Monitoring in Progressive Supranuclear Palsy, an Alzheimer's Disease Related Dementia
Brief Title: Remote Monitoring in Progressive Supranuclear Palsy (PSP)
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Anne-Marie Alexandra Wills, MD, Director, CurePSP Center of Care, Massachusetts General Hospital
Other Study IDs: Not yet available
Record Dates: First submitted 2021-02-06; First posted 2021-02-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Progressive Supranuclear Palsy; Parkinson Disease; MSA - Multiple System Atrophy
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Parkinson Disease; Shy-Drager Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a single-arm, longitudinal, observational study on the use of wearable sensors and digital health technology to measure fall frequency and motor, speech, and cognitive function in patients with PSP over the course of approximately one year. Participants will perform supervised remote assessments monthly and in-person assessments approximately every 6 months.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the feasibility of using wearable sensors and digital health technology to remotely monitor patients with possible or probable PSP.

Secondary objectives are to measure PSP progression using sensor-derived motor and tablet-derived speech and cognitive measures.

In brief, approximately 85 individuals with possible or probable PSP, probable Parkinson's disease, possible or probable Multiple System Atrophy, and healthy controls, will be enrolled at 4-5 sites in the U.S. and followed for one year. During the monitoring period for PSP and MSA participants (1 year), a wearable pendant sensor (PAMSys, BioSensics) will be used to monitor falls and physical activity (step counts) of all participants during activities of daily living (ADL). Parkinson's and healthy control participants will be seen once at baseline only. On a monthly basis, participants will have televideo conferences with the sites to perform supervised gait and balance tasks while wearing 3 LEGSys (BioSensics) sensors. Using a study-supplied tablet, participants will also perform cognitive tests including fluency, color trails and go-no-go tapping tests. Participants will undergo more extensive testing every 3 months including the PSPRS, MoCA, quality of life questionnaires and functional rating scales which will be performed remotely (virtually). Approximately 6 months participants will undergo an in-person PSPRS (to coincide with their clinic appointments).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of possible or probable PSP phenotype as defined by the 2017 MDS criteria, clinical diagnosis of at least probable PD as defined by the 2015 MDS criteria, or clinical diagnosis of at least probable MSA as defined by the 2022 MDS criteria, or healthy controls.
* Male or female, aged 18 to 89 years, inclusive.
* Fluent in reading and speaking English.
* Capable of providing informed consent based on the investigator's judgment.
* Able to comply with the protocol based on the investigator's judgment.
* Able to walk 10 feet unassisted.
* With access to a caregiver who is able to assist with all study-related procedures.

Exclusion Criteria:

* Any neurological, medical, or psychiatric condition that would preclude participation in study activities based on the investigator's judgment.
* A history of frequent falls defined as more than 5 falls/month or requirement of a walker to ambulate safely.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants with clinical diagnosis of possible or probable PSP, probable PD, or possible or probable MSA are eligible to participate in this study. Participants must be able to ambulate unassisted for 10 feet in order to perform gait and balance tests.
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary feasibility outcome | 12 months
  Compliance will be calculated as the number of participants who wear their PAMSys pendant sensors at least 16 hours/day for at least 180 days and complete at least 80% of their scheduled monthly sensor and tablet derived motor, speech, and cognitive assessments through their 6 month visit.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | 12 months
  The Timed Up and Go and other timed gait and balance tests will be performed while wearing LegSys sensors
PSPRS | 12 months
  The Progressive Supranuclear Palsy Rating Scale will be administered remotely or in-person every 3 months. The PSPRS is a 28 item scale with a total score of 0-100 where lower scores are less affected.
MoCA | 12 months
  The Montreal Cognitive Assessment and other cognitive tests will be performed remotely every 3 months. The MoCA is has a total of 30 points and greater than 26 is considered normal.
Cortical Basal ganglia Functional Scale (CBFS) | 12 months
  The Cortical Basal ganglia Functional Scale (CBFS) will be performed every 3 months remotely. The CBFS is a 31 item scale, with a total of 124 possible points, where a lower score is less affected.
PSP-QoL | 12 months
  The PSP Quality of Life scale will be performed every 3 months remotely. The PSP-QoL is a 45 item scale, with a possible scale of 0-100 with lower scores less affected.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie A Wills, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Andrzejewski KL, Dowling AV, Stamler D, Felong TJ, Harris DA, Wong C, Cai H, Reilmann R, Little MA, Gwin JT, Biglan KM, Dorsey ER. Wearable Sensors in Huntington Disease: A Pilot Study. J Huntingtons Dis. 2016 Jun 18;5(2):199-206. doi: 10.3233/JHD-160197. PMID 27341134
- [Background] Raccagni C, Gassner H, Eschlboeck S, Boesch S, Krismer F, Seppi K, Poewe W, Eskofier BM, Winkler J, Wenning G, Klucken J. Sensor-based gait analysis in atypical parkinsonian disorders. Brain Behav. 2018 Jun;8(6):e00977. doi: 10.1002/brb3.977. Epub 2018 May 7. PMID 29733529
- [Background] Espay AJ, Bonato P, Nahab FB, Maetzler W, Dean JM, Klucken J, Eskofier BM, Merola A, Horak F, Lang AE, Reilmann R, Giuffrida J, Nieuwboer A, Horne M, Little MA, Litvan I, Simuni T, Dorsey ER, Burack MA, Kubota K, Kamondi A, Godinho C, Daneault JF, Mitsi G, Krinke L, Hausdorff JM, Bloem BR, Papapetropoulos S; Movement Disorders Society Task Force on Technology. Technology in Parkinson's disease: Challenges and opportunities. Mov Disord. 2016 Sep;31(9):1272-82. doi: 10.1002/mds.26642. Epub 2016 Apr 29. PMID 27125836
- [Derived] Sharma M, Mishra RK, Hall AJ, Casado J, Cole R, Nunes AS, Barchard G, Vaziri A, Pantelyat A, Wills AM. Remote at-home wearable-based gait assessments in Progressive Supranuclear Palsy compared to Parkinson's Disease. BMC Neurol. 2023 Dec 11;23(1):434. doi: 10.1186/s12883-023-03466-2. PMID 38082255